CLINICAL TRIAL: NCT06308328
Title: A Real-world Observational Study of a Mucosal Contouring Method Based on Swallowing-induced Breakthrough Pain for Predicting Radiation-induced Oropharyngeal Mucositis in Patients With Nasopharyngeal Carcinoma
Brief Title: A Real-world Observational Study of a Mucosal Contouring Method for Radiation-induced Oropharyngeal Mucositis
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-090
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Radiation-induced Oropharyngeal Mucositis; Swallowing-induced Breakthrough Pain
Keywords: Nasopharyngeal carcinoma; Radiotherapy; Radiation-induced Oropharyngeal Mucositis; Swallowing-induced Breakthrough Pain; Delineation method
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The performance of the predictive models for the occurrence and severity of oropharyngeal mucositis established using either oral cavity contouring method or mucosa surface contouring method was unsatisfactory in nasopharyngeal carcinoma (NPC). Whereas the predictive model of a mucosal contouring method based on swallowing-induced breakthrough pain exhibited better overall performance in locally advanced NPC. Therefore, the investigators aimed to conduct a prospective, multicenter, real-world observational study to further assess the predictive efficacy of this mucosal delineation method for radiation-induced oropharyngeal mucositis in NPC.

DETAILED DESCRIPTION:
Swallowing-induced breakthrough pain as a prominent clinical challenge for radiation-induced oropharyngeal mucositis, occurs in almost all patients with nasopharyngeal carcinoma (NPC) undergoing radiotherapy, and has a significant impact on patients' quality of life and treatment outcomes. Radiation-induced oropharyngeal mucositis is closely related to the irradiated dose and volume, and the performance of the predictive models for its occurrence and severity established using either oral cavity contouring method or mucosa surface contouring method was unsatisfactory. Thus, it is difficult to carry out risk assessment, precise screening and early intervention through dosimetric parameters, thereby reducing the occurrence of severe radiation-induced oropharyngeal mucositis. The investigators defined a delineation method based on the mucosal areas of radiation-induced injury resulting in swallowing-induced breakthrough pain in locally advanced NPC, and our preliminary results demonstrated that the predictive model exhibited better overall performance. Therefore, the investigators aimed to conduct a prospective, multicenter, real-world observational study to further explore the predictive efficacy of this mucosal delineation method for radiation-induced oropharyngeal mucositis in NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed written consent.
2. Age ≥ 18 years.
3. Histologically confirmed as nasopharyngeal carcinoma, and currently undergoing radical radiotherapy or chemoradiotherapy.
4. Complete and continuous records of oral / oropharyngeal mucositis grading, and self-reported swallowing-induced breakthrough pain.

Exclusion Criteria:

1. Existence of poor oral hygiene, untreated dental or periodontal diseases, and metal dental restorations.
2. Current untreated or unresolved conditions like unstable heart diseases requiring treatment, and poorly controlled diabetes mellitus.
3. Body mass index (BMI) <18.5.
4. Unsuitable to participate in current study, according to researchers' assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with nasopharyngeal carcinoma receiving radical radiotherapy or chemoradiotherapy
Sampling Method: Probability Sample
Enrollment: 718 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The AUC of the predictive model | Through study completion, up to 3 years
  The area under the ROC (receiver operating characteristic) curve (AUC) of the predictive model

SECONDARY OUTCOMES:
The accuracy of the predictive model | Through study completion, up to 3 years
  To obtained this index, true positive (TP) and true negative (TN) were calculated from the confusion matrix.
  Accuracy = (TP+TN)/(Σ Total population)
The sensitivity of the predictive model | Through study completion, up to 3 years
  To obtained this index, true positive (TP) and false negative (FN) were calculated from the confusion matrix.
  Sensitivity = TP/(TP + FN)
The specificity of the predictive model | Through study completion, up to 3 years
  To obtained this index, false positive (FP) and true negative (TN) were calculated from the confusion matrix.
  Specificity = TN/(TN + FP)
The positive predictive value of the predictive model | Through study completion, up to 3 years
  To obtained this index, true positive (TP) and false positive (FP) were calculated from the confusion matrix.
  Positive Predictive value (PPV) = TP/(TP + FP)
The negative predictive value of the predictive model | Through study completion, up to 3 years
  To obtained this index, true negative (TN) and false negative (FN) were calculated from the confusion matrix.
  Negative Predictive value (NPV) = TN/(TN + FN)
The F1 score of the predictive model | Through study completion, up to 3 years
  To obtained this index, true positive (TP), false positive (FP), and false negative (FN) were calculated from the confusion matrix.
  F1 score = 2TP/(2TP + FP + FN)
The important predictors of severe oropharyngeal mucositis in the predictive model | Through study completion, up to 3 years
  The importance of variables included in the predictive model was measure, and those with a higher value indicating a greater contribution to the model's classification accuracy were viewed as the important predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Guan, Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (10):
- China (10):
  - Affiliated Cancer Hospital & Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang hospital, Southern medical university, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Fifth Affiliated Hospital, Sun Yat-sen University, Zhuhai, Guangdong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No